CLINICAL TRIAL: NCT00072644
Title: Pharmacokinetic Interactions With Prednisolone in Healthy Volunteers and HIV-infected Patients Receiving Single-Dose Prednisone
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040040; 04-CC-0040
Record Dates: First submitted 2003-11-06; First posted 2003-11-07 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-06-17

CONDITIONS: Healthy
Keywords: HIV; Osteonecrosis; Drug Interaction; P-Glycoprotein; Cytochrome P 450; Healthy Volunteer; HV
MeSH Terms: conditions — Osteonecrosis

SUMMARY:
This study will evaluate the impact of the HIV protease inhibitor ritonavir on the pharmacokinetics-that is, the interaction of the medication and the body-of prednisolone after prednisone is given to healthy volunteers. Prednisone, an agent known as a corticosteroid, or steroid hormone, is converted by the body into prednisolone. Ritonavir is an HIV medication that fights the virus by blocking its ability to reproduce. Sometimes it increases the blood levels of other drugs given at the same time, and it is possible that ritonavir increases the blood levels of prednisolone and those of other medications. Results from the study will provide information on whether prednisone and ritonavir interact in a potentially harmful way. The MDR1 genotype, that is, part of a person's genetic constitution, may influence how prednisolone behaves.

Patients 18 to 50 years of age who are in good health, who not have HIV, and who do not smoke may be eligible for this study. There will be 10 participants and another 5 later who will be control subjects. Those in the control group will take only prednisone, not ritonavir.

Participants will undergo the following tests and procedures:

* Medical history and physical examination.
* Collection of blood and urine to assess general health.
* Collection of blood to examine markers on white blood cells and to determine the kind of MDR1 gene was inherited.
* HIV test.

The screening visit will take about 3 to 4 hours, and the study will take about 28 to 49 days. For 3 study days, participants will remain in the clinic for 12 hours, On Study Day 1, patients will be asked to not eat or drink anything besides water before coming to the clinic. Blood samples will be collected to measure prednisolone concentration as well as osteocalcin, a blood protein involved in bone formation. Blood tests will also allow a look at the surfaces of some white blood cells. Patients will receive a breakfast along with 20 mg of prednisone. Urine samples will be collected also. Then patients will be dismissed and asked to collect urine samples and return them on the following morning, Study Day 2. At that time there will additional blood collection. Patients will begin taking ritonavir between 7 and 28 days after the first dose of prednisone, at a dose of 200 mg (two 100 mg capsules) twice daily with food, to continue for 15 days. On the 4th and 14th days of their taking ritonavir, patients will be asked to visit the clinic in the morning for a blood to measure ritonavir in the blood and to take a single 20-mg dose of prednisone along with the ritonavir. Both medications will be taken with breakfast. Blood and urine levels of prednisolone will also be measured. On the 15th day of ritonavir dosing, there will be another blood collection for routine lab tests, as well as studies on blood cells and osteocalcin.

DETAILED DESCRIPTION:
Corticosteroid administration has been associated with a variety of toxicities, including osteonecrosis and Cushing's Syndrome, in patients with HIV infection. The prevalence of these toxicities has led to speculation that protease inhibitors impair the cytochrome P450 (CYP) 3A4-mediated metabolism of corticosteroids leading to an increase in their systemic exposure and toxicity. Conversely, reduced corticosteroid exposure may be expected when these drugs are coadministrated with CYP3A4 inducers such as the non-nucleoside reverse transcriptase inhibitor (NNRTI) efavirenz. Despite the hypothesized interaction between antiretroviral medications and corticosteroids, drug interactions between agents from these classes have not been formally investigated. The objectives of this study are (1) to determine the impact of the HIV protease inhibitor ritonavir on the pharmacokinetics of prednisolone after administration of oral prednisone to healthy volunteers and (2) to determine the respective influences of chronic dosing with lopinavir-ritonavir (LPV/r) and efavirenz (EFV) on prednisolone pharmacokinetics in HIV+ individuals taking a single dose of prednisone. For the HIV-negative healthy volunteer portion of the study, 10 HIV-negative study subjects will receive a single 20 mg dose of prednisone before, and after 3 and 14 days of ritonavir exposure at 200 mg twice daily. Blood and urine will be collected over 24 hrs after prednisone administration to determine prednisolone pharmacokinetics and renal elimination. Blood will also be collected for determination of MDR1 genotype, which may influence prednisolone disposition. For the portion of the study conducted in HIV-infected volunteers, 3 groups of 10 subjects will be recruited to receive a single 20 mg dose of prednisone followed by serial blood sampling for prednisolone concentrations. The 3 groups will consist of (1) individuals receiving and HIV treatment regimen (for at least 30 days) that includes LPV/r (2) individuals receiving an HIV treatment regimen (for at least 30 days) that includes EFV and (3) individual receiving no antiretroviral treatment or treatment devoid of HIV protease inhibitors or NNRTIs. Prednisolone concentrations will be determined by validated high performance chromatographic methods. Non-compartmental methods will be used to characterize prednisolone pharmacokinetics in all study groups. Pharmacokinetic parameter values will be compared using ANOVA with post-hoc testing. Geometric mean data with 90% confidence intervals will be reported. This study will characterize, for the first time, the influence of antiretroviral medications on the pharmacokinetics of a corticosteroid medication (prednisolone).

ELIGIBILITY:
* INCLUSION CRITERIA:

HIV-negative Healthy Subjects:

1. Males and females between the ages of 18 and 50 years.
2. Healthy by medical history and physical exam
3. Laboratory values within established guidelines for participation in clinical studies: AST less than or equal to 2 X ULN; Serum creatinine less than or equal to ULN; hemoglobin greater than or equal to 11 g/dL.
4. Ability to abstain from ingesting grapefruit or grapefruit juice during the study period.
5. Negative serum pregnancy test for females of child-bearing potential.
6. Females of child-bearing potential are able and willing to practice abstinence or use non-hormonal effective methods of birth control during the study.
7. Non-smoker for at least 6 weeks prior to study participation.

HIV-infected Volunteers:

1. HIV-infected males and females between the ages of 18 and 50 years.
2. Patients receiving a stable ARV regimen for at least 30 days that includes (1) LPV/r, (2) EFV, or (3) no ARV treatment or treatment that does not contain protease inhibitors, NNRTIs, or other medications known or suspected to alter prednisolone pharmacokinetics.
3. Patients with adequately controlled HIV disease by laboratory and physical exam (HIV-RNA less than 50,000 copies/mL, CD4+ count greater than 200 cells/mm(3), no evidence of active opportunistic infections such as pneumocystis infection, mycobacterial infection etc.)
4. Laboratory values within established guidelines for participation in clinical studies: AST less than or equal to 2X ULN; hemoglobin greater than or equal to 11 g/dL.
5. Ability to abstain from ingesting grapefruit or grapefruit juice for 3 days (2 days before, and the day of prednisone administration).
6. Negative serum pregnancy test for females of child-bearing potential.
7. Females of child-bearing potential are able and willing to practice abstinence or use non hormonal effective methods of birth control during the study.

EXCLUSION CRITERIA:

HIV-negative Healthy Subjects:

1. Concomitant routine therapy with any prescription, over-the-counter, herbal, or holistic medications, including oral contraceptives for 30 days prior to study participation.

   * Subjects must be off oral contraceptives for at least 30 days prior to study day 1.
   * Intermittent (PRN) use of acetaminophen and non-steroidal anti-inflammatory medications (i.e. ibuprofen) will be allowed during the study; these medications should not be taken on days of prednisone administration (study days 1, 10, and 20).
   * Subjects will be allowed to take a multivitamin with minerals, or equivalent, once daily if they desire to do so.
2. Inability to obtain venous access for sample collection.
3. Presence of Diabetes Mellitus, Human immunodeficiency virus (HIV) infection, active tuberculosis, cardiac disease (hypertension; congestive heart failure etc.), renal disease (chronic or acute renal failure or insufficiency), thyroid disease, hepatitis, osteoporosis, osteonecrosis, respiratory disease (asthma requiring chronic treatment; chronic obstructive pulmonary disease), myasthenia gravis, glaucoma, peptic ulcer disease requiring treatment, history of psychiatric illness (other than mild depression or anxiety) or any other condition that may interfere with the interpretation of the study results or not be in the best interest of the subject in the opinion of the investigator.
4. Clinical evidence of adrenal insufficiency, Cushing's Syndrome or any other endocrine disease.
5. Any clinical or laboratory evidence of active infection (persistent fevers, night sweats, nausea, vomiting, diarrhea, chronic cough, WBC greater than the upper limit of normal.)
6. Vaccination within 30 days of study day 1.
7. Exposure to viral illnesses such as chicken pox or measles within 30 days of study participation.
8. Positive pregnancy test or breastfeeding female.
9. The presence of persistent diarrhea or malabsorption that would interfere with the subject's ability to absorb drugs.
10. Drug or alcohol use that may impair safety or adherence.
11. History of intolerance or allergic reaction (rash; hives; swollen lips; difficulty breathing) to corticosteroid medications (e.g. prednisone; prednisolone; methylprednisolone; dexamethasone etc.) or protease inhibitors (ritonavir; lopinavir; amprenavir; indinavir; nelfinavir; saquinavir; atazanavir).
12. Inability or unwillingness of females of child-bearing potential to use a non-hormonal (barrier) method of contraception throughout the study (e.g. condom; diaphragm etc.).
13. Non-fasting total cholesterol or triglycerides greater than or equal to 270 mg/dL.

HIV-infected Volunteers:

1. Concomitant routine therapy with any prescription (including hormonal contraceptives), over-the-counter, herbal, or holistic medications that are known or suspected to alter prednisolone pharmacokinetics.

   * Subjects must be off oral contraceptives for at least 30 days prior to study day 1.
   * Intermittent (PRN) use of acetaminophen and non-steroidal anti-inflammatory medications (i.e. ibuprofen) will be allowed during the study as will vitamin + mineral supplementation.
2. Inability to obtain venous access for sample collection.
3. Patients taking ARV regimens that are not consistent with the study's inclusion criteria; this includes patients taking LPV in combination with EFV or nevirapine.
4. Laboratory and/or physical evidence of any active opportunistic infection.
5. Diabetes Mellitus requiring treatment with oral medications or insulin, active tuberculosis, cardiac disease (uncontrolled hypertension and/or congestive heart failure etc.), renal disease (chronic or acute renal failure or insufficiency resulting in baseline serum creatinine greater than 1.5 X upper limit of normal), untreated/uncontrolled thyroid disease, active hepatitis, respiratory disease (asthma requiring chronic treatment; chronic obstructive pulmonary disease), myasthenia gravis, glaucoma, peptic ulcer disease requiring treatment, history of psychiatric illness (other than mild depression or anxiety) or any other condition that may interfere with the interpretation of the study results or not be in the best interest of the subject in the opinion of the investigator.
6. Clinical evidence of adrenal insufficiency, Cushing's Syndrome or any other endocrine disease.
7. Any clinical or laboratory evidence of active infection (persistent fevers, night sweats, nausea, vomiting, diarrhea, chronic cough, WBC greater than the upper limit of normal.)
8. Vaccination within 30 days of study day 1.
9. Exposure to viral illnesses such as chicken pox or measles within 30 days of study participation.
10. Positive pregnancy test or breastfeeding female.
11. The presence of persistent diarrhea or malabsorption that would interfere with the subject's ability to absorb drugs.
12. Drug or alcohol use that may impair safety or adherence.
13. History of intolerance or allergic reaction (rash; hives; swollen lips; difficulty breathing) to corticosteroid medications (e.g. prednisone; prednisolone; methylprednisolone; dexamethasone etc.).
14. Inability or unwillingness of females of child-bearing potential to use a non-hormonal (barrier) method of contraception throughout the study (e.g. condom; diaphragm etc.).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75
Dates: Start 2003-10-30; Study Completion 2008-06-17

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hammer SM, Squires KE, Hughes MD, Grimes JM, Demeter LM, Currier JS, Eron JJ Jr, Feinberg JE, Balfour HH Jr, Deyton LR, Chodakewitz JA, Fischl MA. A controlled trial of two nucleoside analogues plus indinavir in persons with human immunodeficiency virus infection and CD4 cell counts of 200 per cubic millimeter or less. AIDS Clinical Trials Group 320 Study Team. N Engl J Med. 1997 Sep 11;337(11):725-33. doi: 10.1056/NEJM199709113371101. PMID 9287227